A Prospective Study on the Safety,
Tolerability, and Efficacy of PDR-001
Injection for Bilateral Stereotactic
Subthalamic Nucleus (STN) Clearance of
Alpha-Synuclein

# NIH Clinical Protocol Template: PDR-001 Study

## 1. STUDY OVERVIEW

\*\*Full Protocol Title:\*\*

A Prospective Study on the Safety, Tolerability, and Efficacy of PDR-001 Injection for Bilateral Stereotactic Subthalamic Nucleus (STN) Clearance of Alpha-Synuclein

```
**Protocol ID Number: ** NA
```

## 2. OBJECTIVES AND ENDPOINTS

# 2.1 Primary Objective (52-week Core Phase):

Evaluate the safety and tolerability of PDR-001 injected bilaterally into the STN of patients with early primary PD.

# 2.2 Secondary Objective:

Evaluate the clinical efficacy of PDR-001 within 52 weeks post-injection.

# 2.3 Long-term Objective:

Evaluate long-term safety and efficacy from week 52 up to 5 years.

<sup>\*\*</sup>Version Number and Date:\*\* V1.0, July 6, 2025

<sup>\*\*</sup>Principal Investigator:\*\* Jun Liu

<sup>\*\*</sup>Institution:\*\* Department of Neurology, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine

<sup>\*\*</sup>Study Period:\*\* May 2025 to December 2029

<sup>\*\*</sup>Study Phase:\*\* Phase I/II (Exploratory)

<sup>\*\*</sup>Study Sites:\*\* Single-site trial at Ruijin Hospital, Shanghai

## 2.4 Endpoints

# **Primary Endpoints:**

- Incidence of adverse events (AEs) and serious adverse events (SAEs)
- Change in rAAV neutralizing and binding antibody titers
- Change in whole blood rAAV vector titers

# **Secondary Endpoints:**

- Change in daily Levodopa dose or Levodopa Equivalent Dose (LED)
- Change from baseline in the following scales:
- MDS-UPDRS I-IV
- PGI-I, CGI-I
- MMSE, HAMD, HAMA
- PDSS-2, PDQ-39
- MoCA, NMSQ, SCOPA-AUT, RBDSQ, SS-16, PSQI, Wexner, Berg, Tinetti, Webster, GFQ

# *Long-term Endpoints (52 weeks – 5 years):*

- All primary and secondary endpoints continued over time
- [18F]F-dopa PET gene expression
- DaT-SPECT putaminal binding ratio changes

## 3. BACKGROUND AND RATIONALE

# 3.1 Disease Background

Parkinson's disease (PD) is a progressive neurodegenerative disorder marked by the death of dopaminergic neurons in the substantia nigra. Motor and non-motor symptoms impair

quality of life. In China, PD prevalence ranges from 16.7 to 440.3 per 100,000, affecting 1.7% of the elderly population.

#### 3.2 Unmet Medical Need

Current treatments offer symptomatic relief but do not halt disease progression. Alphasynuclein aggregation is a hallmark of PD pathology. There is a need for innovative therapies that directly target and degrade alpha-synuclein.

# 3.3 Study Agent (PDR-001)

PDR-001 is a novel gene therapy delivered via AAV9 vector encoding a tripeptide (Tat- $\beta$ syndeg) designed to degrade  $\alpha$ -synuclein.

#### 3.4 Preclinical Data

- \*\*Mice (A53T model):\*\* Significant reduction in  $\alpha$ -syn, increased dopaminergic neurons, improved behavior
- \*\*Non-human primates:\*\* Improved motor scores, PET signal in striatum, no systemic toxicity

## 3.5 Rationale for Study Design

First-in-human trial assessing safety and potential clinical benefit of PDR-001 in early-stage PD. Bilateral STN chosen for direct delivery.

#### 3.6 Risk/Benefit Assessment

- \*\*Risks:\*\* Neurosurgical injection, immune response to AAV, transient neuropsychiatric symptoms
- \*\*Benefits:\*\* Potential disease-modifying effect by reducing toxic α-synuclein burden
- \*\*Conclusion:\*\* Favorable risk-benefit ratio supports study initiation

# 4. STUDY DESIGN AND METHODS

#### 4.1 Overall Design

Single-arm, open-label, single-center trial. Total enrollment of 12 participants. Dose-escalation (n=6 in 2 dose levels), followed by an expansion cohort (n=6).

# **4.2 Study Duration**

- 52-week core study
- Up to 5-year long-term follow-up

# 4.3 Sample Size Justification

Exploratory study with 12 patients. No formal power calculation. Safety and biological signals will guide future studies.

# **4.4 Study Intervention**

- \*\*Drug:\*\* PDR-001 injection (AAV9 vector expressing Tat-βsyn-deg)
- \*\*Route: \*\* Bilateral stereotactic injection into the STN
- \*\*Method:\*\* Stereotactic multi-point microinjection (4 targets total)

## 4.5 Study Population

12 patients with early-stage primary PD.

# *Inclusion Criteria (summary):*

- Age 40–65, Hoehn-Yahr ≤ 2, disease duration ≤ 5 years
- Adequate cognitive and liver/renal function
- Negative for HIV, HBV, HCV

## Exclusion Criteria (summary):

- Atypical or secondary Parkinsonism
- History of brain surgery, malignancy, or severe comorbidities

- Pregnancy or nursing

#### **5. STUDY PROCEDURES AND ASSESSMENTS**

Participants will undergo the following evaluations:

- \*\*Preoperative screening:\*\* Informed consent, demographics, physical exam, imaging, lab tests (hematology, biochemistry, serology, pregnancy test), ECG, PD assessments
- \*\*Intervention: \*\* Stereotactic bilateral STN injection of PDR-001 under general anesthesia
- \*\*Follow-up: \*\* At week 4, 12, 26, 39, and 52 post-injection, and every 26 weeks during long-term follow-up. Evaluations include lab tests, imaging (MRI, PET, DaT-SPECT), PD scales, safety assessments

#### 6. SAFETY MONITORING AND ADVERSE EVENT REPORTING

- All AEs and SAEs will be recorded from consent through 52-week core study and throughout long-term follow-up if related to gene therapy.
- SAEs will be reported to the sponsor and Ethics Committee within 24 hours.
- Safety will be reviewed by an independent Safety Review Committee (SRC).

## 7. STATISTICAL ANALYSIS PLAN

- \*\*Descriptive statistics\*\* will summarize safety, tolerability, and efficacy outcomes.
- Categorical data: frequencies and percentages
- Continuous data: mean, median, standard deviation, range
- No formal hypothesis testing due to exploratory nature

#### 8. ETHICAL CONSIDERATIONS

- The study will comply with the Declaration of Helsinki and GCP guidelines.
- Ethics Committee approval is required before initiation.
- Informed consent will be obtained from all participants.

## 9. DATA HANDLING AND RECORD RETENTION

- Electronic Data Capture (EDC) system will be used for data collection.
- All source documents and CRFs will be retained for a minimum of 5 years after study completion.
- Patient confidentiality will be protected through anonymization and restricted access.

# **10. REFERENCES**

(Full reference list available upon request, based on Chinese and international preclinical and clinical gene therapy literature, supporting PDR-001 development.)